CLINICAL TRIAL: NCT00816504
Title: Effect of Galactose on Permeability Factor in Patients With Focal Segmental Glomerulosclerosis (FSGS)and Chronic Kidney Disease Stage 5
Brief Title: Effect of Galactose on Permeblity Factor in Patients With FSGS and CKD Stage 5
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Under additional IRB Review
Sponsor: Northwell Health (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Howard Trachtman MD, Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-124
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: FSGS; Permeability factor; Galactose; Primary FSGS, resistant to immunosuppressive medication
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Galactose
  Interventions: Drug: Galactose

INTERVENTIONS:
Drug: Galactose — Oral galactose, 0.2 g/kg/dose twice daily for 28 days

SUMMARY:
This study is a proof-of-concept clinical study designed to test the hypothesis that oral administration of galactose can lower the level of a circulating factor that increases glomerular permeability to albumin in patients with resistant FSGS.

DETAILED DESCRIPTION:
Patients with resistant FSGS have persistent proteinuria and a high risk of progression to end stage kidney disease (ESKD). A circulating factor that increases glomerular permeability to albumin (Palb) has been detected in over 50% of these patients. While the molecular identity of the factor has not been fully established, in vitro studies and limited clinical experience suggest that galactose can reduce the level of the FSGS permeability factor.

This study is a pilot study to determine if oral administration of galactose can lower the circulating level of the FSGS permeability factor.

Five patients with biopsy proven primary FSGS - native or transplant kidney, receiving plasmapheresis - who are resistant to steroids and one other immunosuppressive agents will be studied.

The only eligibility factor is presence of the FSGS permeability factor.

The experimental intervention is administration of galactose, orally, 0.2 g/kg body weight/dose twice daily. the duration of treatment will be 28 days,.

Patients will be seen on days 0, 14, and 28 of treatment. They will be seen at week 8, 16 and 24 after discontinuation of the galactose.

Physical examination and routine laboratory tests (SMAC, CBC, urine protein:creatinine ratio in an early morning sample) will be done at each visit. The FSGS permeability factor will be assayed at days 0 and 28 of treatment and 6 months after discontinuation of the galactose. The permeability factor will be tested in the laboratory of Virginia Savin MD (Medical college of Wisconsin) using previously described methods.

All other treatments will be unchanged during the 28 day oral galactose Treatment Period.

The study will be analyzed based on the number of patients in whom the FSGS permeability factor is lowered to normal levels.

ELIGIBILITY:
Inclusion Criteria:

* Primary FSGS
* CKD Stage 5
* Resistance to steroids and another immunosuppressive medication

Exclusion Criteria:

* Secondary FSGS

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Reduction in FSGS permeability factor | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — Schneider Children's Hospital
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Trachtman H, Greenbaum LA, McCarthy ET, Sharma M, Gauthier BG, Frank R, Warady B, Savin VJ. Glomerular permeability activity: prevalence and prognostic value in pediatric patients with idiopathic nephrotic syndrome. Am J Kidney Dis. 2004 Oct;44(4):604-10. PMID 15384010